CLINICAL TRIAL: NCT01556828
Title: Analysis of Cutaneous and Hematologic Disorders by High-Throughput Nucleic Acid Sequencing
Status: Terminated | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: LYMNHL0091; SU-03142012-9329 (Other: Stanford University); 21750 (Other: Stanford IRB)
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Cutaneous Lymphoma; Other Skin Disorders; Mycosis Fungoides; Cutaneous T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood tissue
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this study is to identify genetic changes associated with the initiation, progression, and treatment response of response of cutaneous and hematologic disorders using recently developed high-throughput sequencing technologies. The improved understanding of the genetic changes associated with cutaneous and hematologic disorders may lead to improved diagnostic, prognostic and therapeutic options for these disorders.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patient meets the clinical and/or pathologic criteria for the cutaneous or hematologic disorder being examined.
* Patient is willing to provide skin biopsies and five 10 mL tubes of peripheral blood.

Exclusion Criteria:

- Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects will be identified and recruited by referral from that individual's treating physician, mainly Stanford-affiliated dermatologists, oncologists, and hematologists.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2011-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of mutations | 2 years
  Identify mutations, changes in DNA copy number, structural rearrangements, or altered coding and non-coding RNA expression

CONTACTS AND LOCATIONS:
Overall Officials: Paul Khavari, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States